CLINICAL TRIAL: NCT06319196
Title: Clear Me: Interception Trial to Detect and Clear Molecular Residual Disease in Patients With High Risk Melanoma
Brief Title: Clear Me: Interception Trial to Detect and Clear Molecular Residual Disease in Patients With High-risk Melanoma
Acronym: ClearMe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clear Me
Record Dates: First submitted 2024-02-14; First posted 2024-03-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Melanoma; Melanoma Stage IV; Mucosal Melanoma
MeSH Terms: conditions — Melanoma | interventions — Opdualag; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-PD-1/LAG-3 (Opdualag/BMS-986213) (Experimental)
  Interventions: Drug: Opdualag; Drug: Nivolumab
- Anti-PD-1 ( Nivolumab) (Active Comparator)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Opdualag — Opdualag vial IV every 4 weeks (Q4W)
  Other Names: BMS-986213
  Arms: Anti-PD-1/LAG-3 (Opdualag/BMS-986213)
Drug: Nivolumab — Nivolumab 480mg IV Q4W

SUMMARY:
Clear-Me is a biomarker-driven phase II study that tests whether the combination anti- lymphocyte-activation gene-3 (LAG3)/anti-programmed cell death protein 1(PD-1) inhibition Bristol-Myers Squibb (BMS986213) is superior to anti-PD-1 inhibition in patients with detectable circulating tumor deoxyribonucleic acid (ctDNA) following definitive surgery for high risk melanoma. Patients will be allocated to either Arm A or Arm B via the process of randomization. The randomization process will be stratified according to stage (Stage 2A/2B/3A/3B/3C/3D or 4), to ensure absolute balance between stage groups. The investigators are choosing only 1 stratification factor, disease stage, as the investigators consider stage being the most significant prognosticating variable. Each stage represents a biologically distinct entity with varying recurrence rate outcomes. Block randomization will be performed to ensure equal sample sizes in the combination and monotherapy arms. At least 54 patients will be included in the randomized part of the study. The investigators are expecting approximately 20% of the patients to have detectable ctDNA after definite surgery. Therefore, approximately 270 patients are expected to be enrolled and tested for ctDNA in the entire study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening or age of consent according to law.
2. Written informed consent and any locally required authorization (e.g., data privacy) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Must have a life expectancy of at least 12 weeks.
5. Histologically confirmed cutaneous or mucosal melanoma.
6. High risk melanoma subjects with disease staging for which adjuvant immunotherapy has been proven to reduce the risk of relapse versus observation (disease stage: 2B, 2C, 3A, 3B, 3C, 3D, 4 fully resected).
7. Archival tumor formalin-fixed, paraffin-embedded (FFPE) specimens for correlative biomarker studies are required (1 H&E and 10 unstained 5 microns slides). If surgery is going to be performed after signing consent, then tumor FFPE from that surgery is allowed.
8. Patient is a candidate for definitive treatment: including surgery, and post-operative adjuvant immunotherapy with or without radiation for local control.
9. No detectable disease via imaging (CT scan, MRI, with or without Positron emission tomography (PET) CT scan). Table 4.1.2-1 : Criteria for adequate organ and Marrow function
10. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception (see Section 8.1.1 for definition of females of childbearing potential and for a description of highly effective methods of contraception) from screening to 180 days after the final dose of study treatment. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.
11. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from screening to 180 days after receipt of the final dose of study treatment. It is strongly recommended for the female partner of a male subject to also use a highly effective method of contraception throughout this period, as described in Section 8.1.2. In addition, male subjects must refrain from sperm donation while on study and for 180 days after the final dose of study treatment.

Exclusion Criteria:

1. Diagnosis of uveal melanoma.
2. Any prior systemic anticancer therapy for melanoma. Any concurrent anticancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is allowed.
3. Evidence of metastatic disease at surgical and radiological staging.
4. History of allogeneic organ transplantation.
5. History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to anti-PD-1 or anti-LAG-3 or any of their excipients.
6. History of active primary immunodeficiency.
7. Active autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], immune related diverticulitis [prior diverticulitis in the context of diverticulosis is allowed provided is not active], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.].

   The following are exceptions to this criterion:
   1. Participants with vitiligo or alopecia
   2. Participants with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy. Participants without active disease in the last 1 year may be included but only after consultation with the Principal Investigator
   4. Participants with celiac disease controlled by diet alone
8. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive Hepatitis B virus (HBV) surface antigen [HBsAg] result), or hepatitis C (HCV). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with well-controlled Human Immunodeficiency Virus (HIV) are allowed.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, clinically relevant coronary artery disease or history of myocardial infarction in the last 4 months or high risk of uncontrolled arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the participant to give written informed consent.
10. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of study treatment and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
    4. Participants with a history of prostate cancer (tumor/node/metastasis stage) of Stage ≤ T2cN0M0 without biochemical recurrence or progression and who in the opinion of the investigator are not deemed to require active intervention
11. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 500 msecs calculated from three ECGs.
12. Prior nivolumab or relatlimab therapy.
13. Current or prior use of immunosuppressive medication within 14 days before the first dose of study intervention. The following are exceptions to this criterion (see Section 4.7.1.1):

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Participants should not receive live vaccine whilst receiving study intervention and up to 30 days after the last dose of study intervention. Should the participants be deemed candidates for the Monkey pox vaccine, the case will need to be discussed with the coordinating Principal Investigator.
15. Participation in another clinical study with an investigational product administered in the last 28 days prior to randomization or concurrent enrollment in another clinical study, unless the study is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
16. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
17. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
18. Subjects who are unable to willingly provide consent or are unable to comply with the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2030-02-15 (Estimated)

PRIMARY OUTCOMES:
Clearance of ctDNA at 12 months after starting adjuvant treatment. ctDNA clearance is defined as no detection of plasma ctDNA | 12 months after starting adjuvant treatment.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Measured at 12 months and 36 months.
Number and severity of treatment related adverse events according to CTCAE v5.0. | Through study completion, maximum of 6 years.

OTHER OUTCOMES:
Clearance of ctDNA | at month 18 after randomization.
Measured changes of biomarker ctDNA | at 12-week intervals after randomization and up until month 18 after randomization.
Methylation patterns of biomarker ctDNA using circulating free methylated DNA immunoprecipitation and sequencing (cfMeDIPseq) assay and correlation with ctDNA total variant allele frequency (VAF) detection. | Through study completion, maximum of 6 years.
Quality of life assessment using Quality of Life Questionnaire | Performed at pre-dose cycle 1 and 6 (each cycle is 28 days) and end of treatment (within 2 weeks of the subject coming off study therapy)
  patient reported outcomes using 'European Organization for Research and Treatment of Cancer' (EORTC) 'Quality of Life Questionnaire' (QLQ-C30) will be investigated. The score ranges from 1 to 4, with 1 being the worst outcome and 4 being the best. Mean score of individual item numbers of interest will be analyzed with descriptive and mixed effect model methods.

CONTACTS AND LOCATIONS:
Locations (1):
- UHN- Princess Margaret Cancer Center, Toronto, Ontario, Canada